CLINICAL TRIAL: NCT05024188
Title: Assessing the Potential Role of the Gut Microbiome in Modulating Physical Abilities in Humans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf Harofeh MC (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor-Investigator, Assaf Harofeh MC, Principal Investigator, Assaf-Harofeh Medical Center
Organization: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 0277-19-ASF; NCT04707222 (obsolete NCT alias)
Record Dates: First submitted 2021-08-04; First posted 2021-08-27 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Physical Abilities; FMT
MeSH Terms: interventions — Anti-Bacterial Agents; Ciprofloxacin; Metronidazole; Fecal Microbiota Transplantation; Sepharose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotics + FMT (Experimental): 7 days of antibiotics- Ciprofloxacin, 500 mg 2/day & Metronidazole (Flagyl), 500 mg 3/day. After antibiotics administration, participants will receive 10 aFMT capsules for three consecutive days (a total of 30 capsules).
  Interventions: Drug: Antibiotics; Other: Fecal Microbiota Transplantation
- Placebo (Placebo Comparator): 7 days of cellules pills. After cellules pills administration, participants will receive 10 agarose capsules for three consecutive days (a total of 30 capsules).
  Interventions: Other: Cellules Pills; Other: Agarose Capsules

INTERVENTIONS:
Drug: Antibiotics — Ciprofloxacin, 500 mg 2/day & Metronidazole (Flagyl), 500 mg 3/day.
  Other Names: Ciprofloxacin & Metronidazole
  Arms: Antibiotics + FMT
Other: Fecal Microbiota Transplantation — Fecal Microbiota Transplantation is the process of transferring stool from a healthy donor to another.
  Other Names: FMT
  Arms: Antibiotics + FMT
Other: Cellules Pills — 7 days of cellules placebo pills.
  Arms: Placebo
Other: Agarose Capsules — Placebo capsules consist a combination of agarose in normal saline/glycerol (the same vehicle as in a FMT capsules)
  Arms: Placebo

SUMMARY:
The intestinal microbiome is a microbial system that is influenced by host genetics and environmental exposures such as nutrition, stress and medications. There is a growing body of evidence indicating the significant contribution of the gut microbiome to host health and disease. Furthermore, it has been shown that exercise may modify the microbiome composition. However, important mechanistic questions related to the possible associations between exercise and the human gut microbiome remain unanswered.

In this study, the investigators are using advanced state-of-the-art measurements of physical activity level and related metabolic parameters whether there is a connection between the microbiome and physical abilities in healthy participants and whether antibiotics consumption can influence host physical abilities and glycemic responses through changes induced in microbiome composition and function.

DETAILED DESCRIPTION:
During all days of the study, participants will be connected to a continuous glucose monitor (CGM).

In the second segment of the study, participants will be randomized into two groups: antibiotics or placebo, which will be consumed for 7 days.

The third segment of the trial, participants will undergo an FMT/placebo administration for three consecutive days according to their randomization: participants who received antibiotics will receive FMT and participants who received placebo pills will receive placebo capsules in this segment as well.

During the study, participants will collect stool and buccal samples which will be used for microbiota profiling.

Furthermore, participants will undergo physical abilities test, anthropometric measurements, medical history questioners, blood and urine samples and Dual X-ray absorptiometry (DXA) test.

ELIGIBILITY:
Inclusion Criteria:

* BMI<28
* Age - 20-35
* Are used to exercise in aerobic sports (running, swimming, Zumba, ball games, functional training, surfing, tennis, wrestling ext.).
* Exercise at least twice a week, for a minimum duration of the last 6 months.

Exclusion Criteria:

* Consumption of antibiotics (PO) or probiotics 3 months prior to the first day of the experiment.
* Diagnosis of type 1 or type 2 diabetes.
* Pregnancy, fertility treatments, breastfeeding women six months prior to enrollment and during the study.
* Chronic disease (e.g. AIDS, Cushing syndrome, CKD, acromegaly, hyperthyroidism etc.)
* Cancer and recent anticancer treatment
* Psychiatric disorders
* Coagulation disorders
* Gastrointestinal disorders
* Bariatric surgery
* Alcohol or substance abuse
* BMI>28
* Any physical condition precluding the completion of a routine effort test

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-20 (Estimated); Primary Completion 2022-07-20 (Estimated); Study Completion 2023-01-20 (Estimated)

PRIMARY OUTCOMES:
Microbiome Profiling | 2 years
  Collection of stool and buccal samples samples for microbiome composition analysis with16s rRNA sequencing.
Body Mass Index (BMI) | 2 years
  The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m^2
Body Circumferences | 2 years
  waist, hips, and limbs (cm).

SECONDARY OUTCOMES:
Glycemic Responses | 2 years
  Performing continuous glucose monitor (CGM)
Bone Mineral Density (BMD) | 2 years
  Using Dual X-ray absorptiometry (DXA) test

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Youngster, Dr., Principal Investigator — Assaf-Harofeh MC, Bee'r Yaakov Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clarke SF, Murphy EF, O'Sullivan O, Lucey AJ, Humphreys M, Hogan A, Hayes P, O'Reilly M, Jeffery IB, Wood-Martin R, Kerins DM, Quigley E, Ross RP, O'Toole PW, Molloy MG, Falvey E, Shanahan F, Cotter PD. Exercise and associated dietary extremes impact on gut microbial diversity. Gut. 2014 Dec;63(12):1913-20. doi: 10.1136/gutjnl-2013-306541. Epub 2014 Jun 9. PMID 25021423
- [Background] Barton W, Penney NC, Cronin O, Garcia-Perez I, Molloy MG, Holmes E, Shanahan F, Cotter PD, O'Sullivan O. The microbiome of professional athletes differs from that of more sedentary subjects in composition and particularly at the functional metabolic level. Gut. 2018 Apr;67(4):625-633. doi: 10.1136/gutjnl-2016-313627. Epub 2017 Mar 30. PMID 28360096